CLINICAL TRIAL: NCT06718270
Title: A Clinical Study to Explore the Safety, Efficacy, and Pharmacokinetics of CT0596 CAR-T Cell Injection in Patients With Relapsed/Refractory Multiple Myeloma and Relapsed/Refractory Plasma Cell Leukemia
Brief Title: a Study of CT0596 in Relapsed/Refractory Multiple Myeloma and Relapsed/Refractory Plasma Cell Leukemia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT0596-CG6022_01
Record Dates: First submitted 2024-11-24; First posted 2024-12-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-11

CONDITIONS: Relapsed/Refractory Multiple Myeloma; Relapsed/Refractory Plasma Cell Leukemia
Keywords: Relapsed/Refractory Multiple Myeloma; Relapsed or Refractory Plasma Cell Leukemia; CAR-T
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Plasma Cell; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cells Infusion (Experimental): chimeric antigen receptor T cells
  Interventions: Drug: CAR-T cells Infusion

INTERVENTIONS:
Drug: CAR-T cells Infusion — chimeric antigen receptor T cells

SUMMARY:
This study is a single-arm, open-label, exploratory dose-escalation and dose-finding clinical trial to evaluate the safety, efficacy, cellular pharmacokinetics and pharmacodynamics of CT0596 cells in patients with R/R MM and PCL.RRMM and RRpPCL

DETAILED DESCRIPTION:
This study is a single-arm, open-label, exploratory dose-escalation and dose-finding clinical trial to evaluate the safety, efficacy, cellular pharmacokinetics and pharmacodynamics of CT0596 cells in patients with R/R MM and PCL.RRMM and RRpPCL.

During the trial, dose increases or decreases or dose expansion may be performed using i3+3 principle based on the safety and ,tolerability and PK data of the patients.

All Patients will undergo a DLT assessment period which is defined as the first 28 days starting from the day of CT0596 infusion. A patient is evaluable for DLTs if the patient received the planned CT0596 dose and either completed the 28 days of DLT evaluation period after CT0596 infusion or experienced a DLT. Enrolled patients who are not evaluable for DLTs during dose escalation may be replaced. Any Patients who are not DLT evaluable will still be followed for safety and efficacy per the SOA.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be enrolled:

1. Patients must voluntarily sign the informed consent form (ICF) and must be willing and be able to adhere to the trial visit schedule and other protocol requirements and agree to be in long term follow-up (LTFU) for up to 15 years as mandated by the regulatory guidelines.
2. Age ≥ 18 years;
3. Patients with R/RMM who have received at least 3 prior lines of therapy, including at least 1 proteasome inhibitor and at least 1 immunomodulator (IMiD). Patients with RRpPCL had received at least 1 prior line of therapy. Number of lines of therapy was defined according to the guidelines provided in Rajkuma[1]r 2015 . Patients must have received at least 1 complete cycle of therapy for each line of therapy.
4. According to multiple myeloma IMWG 2016 and plasma cell leukemia IMWG 2013, patients must have progressive disease following or during the last treatment.
5. Patients must have measurable disease based on at least one of the following parameters:
6. Expected survival > 12 weeks;
7. Eastern Cooperative Oncology Group (ECOG) score 0- 1 ;
8. Patients should meet the following test results
9. Female patients of childbearing potential must have a negative pregnancy test at screening and prior to receiving lymphodepletion therapy and are willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment and are absolutely prohibited from donating eggs for 1 year after receiving study treatment infusion during the study ;Male patients are willing to use a highly effective and reliable method of contraception for 1 year after receiving study treatment if they are sexually active with a female of childbearing potential. Sperm donation is absolutely prohibited within 1 year following study treatment infusion for all male patients during the study.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patient has any significant condition(s), laboratory abnormality or psychiatric illness that would impair the ability of the patient to receive or tolerate the planned treatment or in the opinion of the investigator, participation would not be in the best interest of the patient (eg, compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
3. Patients seropositive for HIV, active hepatitis C virus (HCV), or active hepatitis B virus (HBV) infection. History of treated hepatitis B or C is permitted if the viral load is undetectable per qPCR and or nucleic acid testing;
4. Patients with any uncontrolled active infection, including but not limited to patients with active tuberculosis (investigator 's judgment);
5. Toxicities caused by previous treatment have not recovered to Common Terminology Criteria for Adverse Events (CTCAE) ≤ Grade 1, except alopecia and other events that are judged tolerable by the investigator;
6. Previous allogeneic stem cell transplantation; autologous stem cell transplantation within 12 weeks prior to signing informed consent;
7. Have received treatment for the disease within 14 days before informed consent
8. Have received cell therapy within 28 days before informed consent.
9. Systemic glucocorticoids equivalent to > 15 mg/day prednisone within 7 days prior to informed consent, with the exception of topical glucocorticoids;
10. Vaccination with live attenuated vaccines , inactivated vaccines or RNA vaccines within 4 weeks prior to informed consent;
11. Allergic or intolerant to lymphodepletion, tocilizumab, or allergic to components (DMSO) in CT0596 CART cell infusion preparation; or previous history of other serious allergies such as anaphylactic shock;
12. Patients Waldenström macroglobulinemia, POEMS syndrome, or primary light chain amyloidosis at Screening;
13. Patients with any of the following cardiac conditions within 6 months prior to screening:
14. Patients who require supplemental oxygen to maintain oxygen saturation > 92%; or Patients with known or suspected COPD who have Forced Expiratory Volume in 1 second (FEV1) < 50% of predicted normal on spirometry;
15. Patients with active autoimmune diseases, including but not limited to psoriasis, rheumatoid arthritis and other diseases requiring long-term immunosuppressive therapy;
16. Patients with second primary malignancies are not eligible if the second primary malignancy has required treatment within the past 2 years or is not in complete remission. Exceptions include the following that have been successfully treated - nonmetastatic basal cell or squamous cell skin carcinoma, non-metastatic prostate cancer, carcinoma-in-situ of breast or cervix, non-muscle invasive bladder cancer
17. Patients with symptomatic central nervous system (CNS) disease or suspected CNS metastases;
18. Major surgery within 2 weeks before informed consent or planned during the study period or within 4 weeks after giving study treatment (excluding local anesthesia such as cataract)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2027-01-03 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AE) after CT0596 infusion | 12 months after CT0596 infusion
  An assessment of severity grade will be made according to the National Cancer Institute Common Terminology Criteria
MTD and/or dose range | 12 months after CT0596 infusion
  Evaluate Dose limited toxicity and recommended dosage range after CT0596 infusion

SECONDARY OUTCOMES:
Overall response rate (ORR) as assessed by the investigator | 12 months after CT0596 infusion
  Overall response rate (ORR) defined as proportion of patients achieving partial response or better based on International Myeloma Working Group defined response criteria
Complete response/stringent complete response (CR/sCR) rate | 12 months after CT0596 infusion
  Rate of complete response/stringent complete response (CR/sCR) defined as proportion of patients achieving CR or better based on IMWG defined response criteria.
Rate of very good partial response (VGPR) and above | 12 months after CT0596 infusion
  Rate of complete very good partial response response/stringent complete response (VGPR/CR/sCR) defined as proportion of patients achieving VGPR or better based on IMWG defined response criteria
Duration of response (DOR) | 12 months after CT0596 infusion
  DOR is defined as the time from first achieving PR or better to confirmed disease progression or death from any cause
Minimal residual disease (MRD) negative rate | 12 months after CT0596 infusion
  Minimal residual disease (MRD) negative rate is defined as the proportion of patients with VGPR or better who achieved 10-5 sensitivity of nucleated cell
Time to response (TTR) | 12 months after CT0596 infusion
  TTR defined as the time from the date of apheresis to the date of initial assessment of PR or better according to IMWG2016 criteria
Progression-free survival (PFS) | 12 months after CT0596 infusion
  PFS defined as the time from the date of apheresis of the subject to the first assessment of confirmed disease progression or death from any cause according to IMWG2016 criteria, whichever occurs first.
Peak value of CART cells | 12 months after CT0596 infusion
  Time to peak expansion and peak expansion in plasma after infusion of CT0596 cells
Overall survival (OS) | 12 months after CT0596 infusion
  OS defined as the time from the date of apheresis of the subject to death from any cause
Cytokines in the peripheral blood after CT0596 infusion | 12 months after CT0596 infusion
  Serum concentrations of interleukin (IL)-6 after CT0596 infusion
Area under the plasma concentration versus time curve (AUC) of CART cells | 12 months after CT0596 infusion
  Area under the plasma concentration versus time curve (AUC) in plasma after infusion of CT0596 cells
In vivo persistence of CART cells | 12 months after CT0596 infusion
  CART cells duration in plasma after infusion of CT0596 cells

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, Ph D, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China